CLINICAL TRIAL: NCT00729963
Title: Efficacy of Sibutramine-induced Weight Loss vs. Continuous Positive Airway Pressure (CPAP) in the Treatment of Obese Patients With Obstructive Sleep Apnea
Brief Title: Sibutramine Versus Continuous Positive Airway Pressure (CPAP)in Obstructive Sleep Apnea (OSA) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Frédéric Sériès, Laval Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CER911
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Obstructive Sleep Apnea; Obesity; Hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Hypertension | interventions — sibutramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The first group received sibutramine 10 mg for the first 4 weeks, at which time consideration of increasing dosage to 15 mg was re-evaluated in the case of insufficient weight loss (< 1.8 kg) over the first month of treatment.
  Interventions: Drug: Sibutramine
- 2 (Active Comparator): A standard reference group, which was paired according to age and BMI, received CPAP as a treatment for OSA.
  Interventions: Device: CPAP

INTERVENTIONS:
Drug: Sibutramine — The first group received sibutramine 10 mg for the first 4 weeks, at which time consideration of increasing dosage to 15 mg was re-evaluated in the case of insufficient weight loss (< 1.8 kg) over the first month of treatment.
  Arms: 1
Device: CPAP
  Arms: 2

SUMMARY:
The primary objective of this study is to observe if Sibutramine is effective in improving the symptoms and signs of sleep apnea in obese patients. The secondary objectives are to document the effects of Sibutramine on heart rate variability and 24-h arterial pressure values. We hypothesized that sibutramine will improve sleep disordered breathing, cardiac autonomic function and systemic blood pressure in obese patients with obstructive sleep apnea (OSA).

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants with non-treated OSA syndrome were aged between 18 to 65 years, with a body-mass index (BMI) ≥ 30 kg/m2 or ≥ 27 kg/m2 in the presence of other risk factors such as controlled systemic hypertension, type 2 diabetes, dyslipidemia and/or visceral obesity (as defined by a waist circumference ≥ 102 cm in men and ≥ 88 cm in women).

Exclusion Criteria:

* Exclusion criteria were uncontrolled systemic hypertension defined as blood pressure > 145/90 mm Hg, previous pharmacological or surgical treatment for weight loss, had already used CPAP or had severe diurnal hyper somnolence requiring immediate treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

REFERENCES:
- [Derived] Ferland A, Poirier P, Series F. Sibutramine versus continuous positive airway pressure in obese obstructive sleep apnoea patients. Eur Respir J. 2009 Sep;34(3):694-701. doi: 10.1183/09031936.00167308. Epub 2009 Apr 8. PMID 19357147